CLINICAL TRIAL: NCT03273764
Title: Development And Validation Of A Clinical RD Score For Decision Making For Administration Of Surfactant In Preterm Babies With RDS (Respiratory Distress Syndrome) - A Prospective Observational Study
Brief Title: Clinical RD (Respiratory Distress) Score for Objective Decision Making for Surfactant Therapy
Status: Completed | Type: Observational
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Director professor and head of department, Lady Hardinge Medical College
Other Study IDs: LadyHardingeMedicalCollege
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Surfactant; CPAP
Keywords: Preterm, RDS, Surfactant, CPAP
MeSH Terms: conditions — Premature Birth; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm neonates with RDS: Singleton Preterm neonates with gestational age between 26 completed weeks to 34 completed weeks with clinical diagnosis of RDS without any major congenital anomalies.

SUMMARY:
To develop a comprehensive 'Clinical RD score' for decision making for administration of Surfactant in respiratory distress syndrome in preterm infants with gestation of 26 0/7 - 34 6/7 weeks and to assess the validity of this 'clinical RD score' on a different subgroup of patients with similar gestational age.

DETAILED DESCRIPTION:
Respiratory distress syndrome, also known as hyaline membrane disease, occurs almost exclusively in premature infants. The incidence and severity of respiratory distress syndrome are inversely related to the gestational age of the newborn infant. The incidence of RDS is around 60 - 80% among infants < 28 weeks, 30-40% between 28-34 weeks, less than 5% at 34 weeks and is rarely seen among those > 37 weeks.

The availability of continuous positive airway pressure (CPAP) and natural surfactant have revolutionised the management of RDS. In 1967, Gregory et al. reported the value of application of continuous positive airway pressure in the management of RDS. Successful surfactant replacement therapy in RDS was reported by Fujiwara et al. Besides the use of Continuous positive airway pressure and surfactant replacement, the other advances include: Use of antenatal steroids to enhance pulmonary maturity, appropriate resuscitation and immediate use of CPAP for alveolar recruitment, Use of gentler modes of ventilation like patient triggered ventilation, Supportive therapies, such as the diagnosis and management of patent ductus arteriosus (PDA), fluid and electrolyte management, trophic feeding and nutrition.

The use of CPAP applied to the alveoli has been shown to stabilise and improve respiratory distress in preterm babies. It preserves the action of endogenous surfactant and may also obviate the need for surfactant in a substantial number of cases. CPAP is cost effective and more patient friendly than mechanical ventilation. Availability of CPAP even at the district level Special Newborn Care Unit (SNCU) in various states across the country make it an ideal candidate for respiratory support in the high risk population.

In addition to optimal respiratory support in the form of continuous positive airway pressure (CPAP) or mechanical ventilation and good supportive care, surfactant replacement therapy (SRT) forms the mainstay in the management of RDS. Since the report by Fujiwara in 1980 of the first successful use of SRT, numerous randomized controlled trials (RCTs) and their meta-analyses have established its efficacy in reducing mortality and air leak syndromes in RDS. Almost all the trials evaluating the role of SRT were conducted in high-income countries. Not surprisingly, SRT is the standard of care in neonates with RDS in these countries.

The population in low and middle income countries (LMIC) like India may differ significantly from the western world. But whether the evidence from these high income countries can be extrapolated to LMICs, still remains questionable. High cost of surfactant therapy, issue regarding regular supply of the drug, lack of skilled personnel, poor antenatal steroid coverage of mothers with preterm labour, higher incidence of perinatal hypoxia/ischemia and infections all complicate the clinical course of RDS. The paucity of evidence for efficacy and/ or safety of SRT in these settings further add to the complexity.

Continuous positive airway pressure (CPAP) remains as the first line of respiratory support in spontaneously breathing infants with RDS and surfactant is administered if required. The beneficial effects of surfactant are more pronounced when the therapy is started earlier. In most of the units across the country, the decision to administer surfactant to such babies managed on CPAP is clinician oriented and hence remains highly subjective. There are no objective criteria to decide for administration of surfactant to infants who are initially managed with CPAP. The current study was planned keeping in mind the beneficial effects of early CPAP and early surfactant, with the aim of developing an objective scoring system, which would guide the clinician in decision making for administration of surfactant to infants with RDS who are already being managed with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Neonates between 26 0/7-34 6/7 weeks of gestation who were delivered in the hospital with clinical diagnosis of respiratory distress syndrome were eligible for inclusion for the study.

Exclusion Criteria:

* Major congenital malformation
* Antenatally diagnosed congenital heart disease in fetus.
* Hydrops fetalis
* Massive Pulmonary hemorrhage prior to enrolment
* Shock requiring vasopressor support prior to enrolment
* Non availability of CPAP/ventilator in the unit.

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates between 26 weeks to 34 weeks of gestation with a clinical diagnosis of RDS.
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Developement of a clinical RD score for decision making for administration of surfactant in preterm babies with RDS | January 2015 to September 2016
  The study will be conducted in 2 parts.Written informed consent will be obtained from one of the parents of the eligible neonates. The demographic and clinical data related to all putative risk factors will be recorded at the time of enrollment from all eligible neonates in the age group of 26-34 weeks with clinical features suggestive of RDS/HMD (Hyaline Membrane Disease). The putative risk factors which could potentially increase the chances of surfactant administration to the infant will be documented and will be analysed through logistic regression analysis and clinical RD score will be developed. The score developed in the first part of the study will be applied on a different population of preterm infants with RDS with similar gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Principal Investigator — Kalawati Saran Chindren Hospital and Lady Hardinge Medical College; Debasish Nanda, MBBS, MD, Principal Investigator — Kalawati Saran Chindren Hospital and Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical college, New Delhi, National Capital Territory of Delhi, India